CLINICAL TRIAL: NCT06628765
Title: Two Types of Single-use Flexible Ureteroscopies for the Treatment of Upper Urinary Tract Stones in Children: A Single-center Randomized Controlled Trial
Brief Title: Two Types of Single-use Flexible Ureteroscopies for the Treatment of Upper Urinary Tract Stones in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Hongbo Liu, Principal Investigator, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-IRB-0310-P-01
Record Dates: First submitted 2024-09-28; First posted 2024-10-08 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Urinary Stone
Keywords: Urinary Stone; Flexible Ureteroscopy; Children
MeSH Terms: conditions — Urinary Calculi

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 8.6 Fr single-use fURS (XFGC-FU-660RC) (Active Comparator): 8.6 Fr single-use fURS (XFGC-FU-660RC) arm received 8.6 Fr single-use fURS
  Interventions: Device: 8.6 Fr single-use fURS (XFGC-FU-660RC)
- 6.3 Fr single-use fURS (HugeMed, HU30S) (Experimental): 6.3 Fr single-use fURS (HugeMed, HU30S) arm received 6.3 Fr single-use fURS
  Interventions: Device: 6.3 Fr single-use fURS (Hugemed, HU30S)

INTERVENTIONS:
Device: 8.6 Fr single-use fURS (XFGC-FU-660RC) — Comparative device
  Arms: 8.6 Fr single-use fURS (XFGC-FU-660RC)
Device: 6.3 Fr single-use fURS (Hugemed, HU30S) — Device being tested
  Arms: 6.3 Fr single-use fURS (HugeMed, HU30S)

SUMMARY:
The single-use digital flexible Ureteroscopy (fURS) is commonly used for the treatment of upper urinary tract stones. The size of the outer diameter of the fURS can affect the safety, efficacy, and medical costs of the treatment. Particularly for children, their ureters are thinner and more tortuous compared to adults, which places higher demands on medical devices. The investigators are interested in determining if the performance of the two different sizes of fURS (6.3 Fr vs. 8.6 Fr) are equivalent. This study will have guiding significance for the selection of upper urinary tract stones surgery in children in the future.

DETAILED DESCRIPTION:
The single-use digital fURS is a sterile, disposable, flexible endoscope. Compared to traditional reusable digital flexible endoscopes, single-use digital fURS has lower maintenance costs, is easier to operate, and effectively avoids cross-infection between patients. With technological advancements, the size of single-use digital fURS has become increasingly slim, making them particularly suitable for children with narrow and tortuous ureters who suffered urinary stones. Currently, the single-use digital fURS used in our unit has an outer diameter of 8.6Fr. For younger children, the success rate of the first insertion of the fURS is still relatively low. When the fURS cannot pass through the ureter, it is necessary to actively dilate the ureter with a balloon in one stage, or passively dilate it with a urethral stent during the procedure to facilitate a second-stage fURS procedure. This not only increases the risk of ureteral injury but also incurs additional medical expenses. Recently, HugeMed Company has launched a single-use digital fURS with an outer diameter of 6.3 Fr, which is currently the thinnest single-use fURS in the world, and its effectiveness and safety have been preliminarily verified in clinical practice. The purpose of this study is to compare the safety and efficacy of the 6.3 Fr fURS (HU30S) and the 8.6 Fr fURS (XFGC-FU-660RC) in the clinical treatment of upper urinary tract stones in children.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for ureteroscopy and laser lithotripsy for individual renal stones ranging in size from 5 mm to 20 mm in all intrarenal locations (If there are multiple stones present, the total stone burden in cross section should not exceed 20 mm)
* Patients < 14 years
* For children younger than 8 years old, the informed consent form is signed by the parents; for children older than 8 years old, the informed consent form is signed by both the parents and the child themselves.

Exclusion Criteria:

* Children with uncontrolled urinary tract infections or coagulation disorders and other contraindications for surgery before the operation.
* Children with severe renal insufficiency, anatomical or functional solitary kidney, known nephrocalcinosis, and other significant comorbidities that are not suitable for participating in the study.
* Children who refuse to participate in this study.
* Any other reason that in the opinion of the investigator would make the participant unsuitable for enrollment in the study.

Ages: 0 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-04-08 (Estimated); Study Completion 2025-04-08 (Estimated)

PRIMARY OUTCOMES:
The success rate of the first fURS insertion | During the procedure
  The first insertion of fURS is successful without the need for balloon dilation or passive dilation with a stent.

SECONDARY OUTCOMES:
Ureteral access sheath placement (Yes/No) | During the procedure
  Whether a ureteral access sheath is placed during the procedure
Balloon dilation rate | During the procedure
  Due to difficulty in passing the fURS through the ureter, balloon dilation of the ureter is performed during the procedure
Pre-placement rate of double-J stents | During the procedure
  Due to difficulty in passing the fURS through the ureter, the double-J stent is placed during the surgery to passively dilate the ureter, facilitating a second-stage fURS procedure
Surgical duration | During the procedure
  From the initiation of fURS insertion to the completion of lithotripsy, the fURS is withdrawn from the body
Blood loss | During the procedure
  Intraoperative blood loss
Indwelling catheter duration | Three days postoperatively
  Indwelling catheter duration postoperatively
Postoperative hospital stay | Up to one week postoperatively
  Postoperative hospital stay
Perioperative complications | Through study completion, up to two months postoperatively
  Pain (e.g. dysuria and lumbar pain), Hematuria, Frequency and urgency of urination, Fever
Stone-free rate at 4 weeks postoperatively | 4 weeks postoperatively
  Stone-free status was evaluated at 4-week and defined as a single residual fragment ≤2 mm

CONTACTS AND LOCATIONS:
Overall Officials: Hongbo Liu, Principal Investigator — Children's Hospital, Zhejiang University School of Medicine
Locations (1):
- Children's hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China